CLINICAL TRIAL: NCT02028871
Title: Intranasal Insulin for Weight Management During Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajna Hamidovic (Other)
Responsible Party: Sponsor-Investigator, Ajna Hamidovic, Assistant Professor, University of New Mexico
Organization: University of New Mexico (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 120700
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Tobacco Abstinence Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Insulin First (Active Comparator): Intranasal Insulin First, Placebo Second
  Interventions: Drug: Intranasal Insulin
- Placebo First (Placebo Comparator): Placebo First, Intranasal Insulin Second
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Insulin
  Arms: Intranasal Insulin First
Drug: Placebo
  Arms: Placebo First

SUMMARY:
This FDA-approved (IND# 120700) study will evaluate efficacy of intranasal insulin in reducing snack intake and reducing postprandial free fatty acid levels in abstinent smokers.

ELIGIBILITY:
Inclusion Criteria:

* smokers (>10 cig/day) for the past 1 year
* normosmic olfactory function

Exclusion Criteria:

* previous/current use of insulin
* current Diagnostic and Statistical Manual-IV-Revised (DSM-IV-R) Axis I disorder
* current pregnancy (or lactation)
* lifetime history of endocrine disease
* excessive alcohol use (>25 standard units of alcohol/week)
* current use of illicit drugs
* current use of a smoking cessation aid (NRT, Chantix or Wellbutrin), or a psychotropic agent
* local infections, inflammation, structural abnormalities, or other nasal pathology
* current use of any medications administered intranasally, including intranasal steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajna Hamidovic, PharmD, Principal Investigator — University of New Mexico
Locations (1):
- UNM College of Pharmacy, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Insulin Arm: Active Treatment First
- Placebo: Placebo treatment first
Period: Overall Study
Arm/Group | Intranasal Insulin Arm | Placebo
Started | 14 | 12
Completed | 10 | 9
Not Completed | 4 | 3
Not completed — Positive urine drug screen | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — IV placement difficulty | 1 | 0
Not completed — Current Illness | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo first
- Total: Total of all reporting groups
Arm/Group | Placebo | Intranasal Insulin Arm | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.33 (12.82) | 29.30 (7.14) | 33.57895 (10.81198)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 9 | 13
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Amount Eaten in Taste Test
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Intranasal Insulin Arm: Active Treatment
- Placebo: Placebo treatment
Arm/Group | Intranasal Insulin Arm | Placebo
Number analyzed (Participants) | 19 | 19
grams | 124 (48) | 116 (66)

2. Other Pre Specified Outcome: Nicotine Cravings Measured by Questionnaire of Smoking Urges
Description: Range: 7-70. Higher scores mean worse outcome
Time Frame: 210 minutes
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Placebo
Arm/Group | Placebo | Intranasal Insulin Arm
Number analyzed (Participants) | 19 | 19
score on a scale | 35.98 (1.20) | 32.52 (1.05)

ADVERSE EVENTS:
Time Frame: 240 minutes
Groups:
- Intranasal Insulin: Group Receiving Intranasal Insulin
- Placebo: Group Receiving Placebo
- Follow up: Total Participants Completed Study
Arm/Group | Intranasal Insulin | Placebo | Follow up
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/19
Other Adverse Events (participants affected / at risk) | 11/26 | 7/24 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Insulin (N=26) | Placebo (N=24) | Follow up (N=19)
Irritation (General disorders) | 5 (7) | 3 (5) | 1 (1) — Nasal Occurrences
Dizziness (General disorders) | 1 (1) | 0 (0) | 1 (1) — Other Occurrences
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) — Other Occurrences
Confusion (General disorders) | 2 (2) | 1 (1) | 0 (0) — Other Occurrences
Tingling (mouth) (General disorders) | 1 (1) | 0 (0) | 0 (0) — Other Occurrences
Shaking (General disorders) | 1 (1) | 0 (0) | 1 (1) — Other Occurrences
Smell (General disorders) | 1 (2) | 1 (1) | 0 (0) — Nasal Occurrences
Sneezing (General disorders) | 1 (2) | 1 (1) | 0 (0) — Nasal Occurrences
Congestion (General disorders) | 1 (2) | 2 (3) | 0 (0) — Nasal Occurrences
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Nasal Occurrences
Fainter Sniffin Sticks (General disorders) | 2 (2) | 0 (0) | 1 (1) — Nasal Occurrences
Nasal Abrasions (General disorders) | 1 (1) | 0 (0) | 0 (0) — Nasal Occurrences
Sweating (General disorders) | 2 (2) | 0 (0) | 0 (0) — Other Occurrences
Visual Disturbances (General disorders) | 0 (0) | 0 (0) | 1 (1) — Other Occurrences
Anxiety (General disorders) | 1 (1) | 1 (1) | 0 (0) — Other Occurrences
Itchiness (General disorders) | 0 (0) | 0 (0) | 0 (0) — Other Occurrences
Diarrhea (General disorders) | 0 (0) | 0 (0) | 1 (1) — Other Occurrences
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) — Other Occurrences
Body Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Other Occurrences
Menorrhagia (General disorders) | 0 (0) | 0 (0) | 1 (1) — Other Occurrences
Restlessness (General disorders) | 1 (1) | 0 (0) | 0 (0) — Other Occurrences
Confined (General disorders) | 1 (1) | 0 (0) | 0 (0) — Other Occurrences
Uncomfortable (General disorders) | 1 (1) | 0 (0) | 0 (0) — Other Occurrences
Eyes Watering (General disorders) | 1 (2) | 1 (1) | 0 (0) — Other Occurrences
Hunger (General disorders) | 1 (1) | 1 (1) | 0 (0) — Other Occurrences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes